CLINICAL TRIAL: NCT02326922
Title: The Use of Levonorgestrel-Releasing Device (Metraplant-E) in the Treatment of Dysfunctional Uterine Bleeding
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmad Aboulfetouh Mahmoud, Obgyn resident, Ain Shams Maternity Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAM1983
Record Dates: First submitted 2014-06-29; First posted 2014-12-30 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Dysfunctional Uterine Bleeding
Keywords: Dysfunctional uterine bleeding; Metraplant-E; Levonorgestrel-releasing intrauterine device; Endometrial decidualization
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metraplant-E First prototype (Experimental): Metraplant-E (first prototype) levonorgestrel-releasing intrauterine device
  Interventions: Device: Metraplant-E levonorgestrel-releasing intrauterine device
- Metraplant-E second prototype (Experimental): Metraplant-E (second prototype) levonorgestrel-releasing intrauterine device
  Interventions: Device: Metraplant-E levonorgestrel-releasing intrauterine device

INTERVENTIONS:
Device: Metraplant-E levonorgestrel-releasing intrauterine device — Metraplant-E insertion and follow up for 6 months

SUMMARY:
Research hypothesis: Release of levonorgestrel from Metraplant-E levonorgestrel releasing intrauterine contraceptive device is inadequate to be used as a medical line of treatment of dysfunctional uterine bleeding.

The investigators aim to evaluate the therapeutic effect of the intrauterine system (Metraplant-E) in the treatment of dysfunctional uterine bleeding.

DETAILED DESCRIPTION:
Primary outcome : The investigators aim to evaluate the short term release of levonorgestrel from the Metraplant-E levonorgestrel releasing intrauterine contraceptive devices (IUCDs). This is in a trial to determine to what extent the intrauterine release of levonorgestrel would reduce MBL in women with menorrhagia and if the treatment would increase the body iron stores and the degree of patient satisfaction and acceptability of treatment for the patients with dysfunctional uterine bleeding. This will be conducted through a questionnaire offered to the women participating in this study which is designed on Likert scale.

Secondary outcome:

1) Endometrial biopsy prior to and 6 months after the insertion of the intrauterine system (Metraplant-E).

3) Haemoglobin level measurement in gm/dl and serum ferritin level on same occasions as when endometrial biopsy is done.

4) The amount of monthly menstrual blood loss after the insertion the Metraplant-E levonorgestrel releasing intrauterine contraceptive devices using the following scores: bleeding index,total bleeding score and Pictorial blood loss assessment chart (PBAC).

Inclusion criteria:

1. Women seeking contraception.
2. Women with history of menorrhagia.
3. Pre and perimenopausal women who are married or previously married.
4. Failure of other medical treatment to control menorrhagia such as hemostatics.
5. Women who did not tolerate copper IUD (intrauterine device) due to increased amount of menstrual blood loss which could lead to anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Women seeking contraception.
2. Women with history of menorrhagia.
3. Pre and perimenopausal women who are married or previously married.
4. Failure of other medical treatment to control menorrhagia such as hemostatics.
5. Women who did not tolerate copper IUD due to increased amount of menstrual blood loss which could lead to anemia.

Exclusion Criteria:

1. History of ectopic pregnancy .
2. Pregnancy or suspicion of pregnancy.
3. Congenital or acquired uterine anomaly including fibroids if they distort the uterine cavity.
4. Acute pelvic inflammatory disease
5. Postpartum endometritis or infected abortion in the past 3 months.
6. Known or suspected uterine or cervical neoplasia or unresolved, abnormal Pap smear.
7. Genital bleeding of unknown etiology.
8. Untreated acute cervicitis or vaginitis, including bacterial vaginosis or other lower genital tract infections, until infection is controlled.
9. Acute liver disease or liver tumor (benign or malignant).
10. Conditions associated with increased susceptibility to infections with microorganisms. Such conditions include, but are not limited to, leukemia, acquired immune deficiency syndrome (AIDS), and I.V. drug abuse.
11. A previously inserted IUD that has not been removed.
12. Hypersensitivity to any component of this product.
13. Women taking anticoagulants
14. Women with coagulopathies due to thrombocytopenia or platelets dysfunction.
15. Known or suspected carcinoma of the breast.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Amount of menstrual blood loss (MBL) in women with menorrhagia by means of pictorial bleeding assesment chart | 6 months
  This is in a trial to determine to what extent the intrauterine release of levonorgestrel would reduce menstrual blood loss (MBL) in women with menorrhagia and if the treatment would increase the body iron stores and the degree of patient satisfaction and acceptability of treatment for the patients with dysfunctional uterine bleeding. This will be conducted through a questionnaire offered to the women participating in this study which is designed on Likert scale.

SECONDARY OUTCOMES:
Histological changes in Endometrial biopsy prior to and 6 months after the insertion of the intrauterine system (Metraplant-E) | 6 months
  to observe the effects of the intrauterine-released levonorgestrel on the endometrium after 6 months after the insertion of the device
Hemoglobin level in blood prior to the device insertion and 6 months afterwards | 6 months
  and to assess the effect on general condition of the patient by following up the haemoglobin level.

OTHER OUTCOMES:
The degree of patient satisfaction and acceptability of treatment Metraplant-E intrauterine device for the patients with dysfunctional uterine bleeding. | 6 months
  This will be conducted through a questionnaire offered to the women participating in this study which is designed on Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Azzam, MD, Study Director — Ain Shams University Faculty of Medicine
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided